CLINICAL TRIAL: NCT04359706
Title: Bacterial and Fungal Microbiota of Patients With Severe Viral Pneumonia With SARS-CoV2
Brief Title: Bacterial and Fungal Microbiota of Patients With Severe Viral Pneumonia With COVID-19
Acronym: MICROVID
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_28; 2020-A01042-37 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2020-04

CONDITIONS: Sars-CoV2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bronchoalveolar lavage and rectal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid-19 group: Critically ill patients with SARS-CoV-2 infection
- control group: Historical critically ill patients with no SARS-CoV-2 infection

SUMMARY:
Observational pilot single-center study aiming to determine the microbiota of critically ill patients infected with SARS-CoV-2. COVID-19 patients will be compared to historical critically ill controls with no SARS-CoV-2 infection.

DETAILED DESCRIPTION:
Observational pilot single-center study aiming to determine the microbiota of critically ill patients infected with SARS-CoV-2. COVID-19 patients will be compared to historical critically ill controls with no SARS-CoV-2 infection.

Respiratory and fecal microbiota (microbial and fungal) will be determined in COVID-19 patients on bronchoalveolar lavage and rectal swab.

Inflammatory biomarkers will also be measured in COVID-19 patients.

Characteristics of study patients will be collected at ICU admission and during ICU stay.

ELIGIBILITY:
Inclusion Criteria:

For the Covid-19 Group: with a confirmed severe lung infection with CoV2-SARS-Cov2 admitted to the ICU.

For the Control Group:

* Historic cohort of non SARS -CoV2-infected adults admitted to the ICU (between March and October 2019),
* that was investigated for fecal microbiota in a previous study (control patients in a fecal microbiota study in patients included in the SEAT study).

Exclusion Criteria:

* For the Covid-19 group:
* Lack of coverage Patients who received antibiotic therapy within 6 weeks prior to Covid-19 symptomatology,
* Pregnant women,
* Severe immunosuppression: Neutropenia < 0.5 G/L, Chemotherapy < 6 months, Bone marrow transplant recipients, HIV with CD4+ lymphocytes < 0.4 G/L
* Impossible to perform bronchoalveolar lavage,
* Non-socially insured,
* Refusal to participate in the social study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients suspected of SARS-CoV2 infection and admitted in ICU
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Composition of the fecal bacterial and fungal microbiota | At 28 days
  relative abundances and diversity indices

SECONDARY OUTCOMES:
Analysis of the faecal microbiota from rectal swab | at baseline and every 7 days during 28 days
  Alterations in fecal microbiota composition (including virose, bacteria and fungi) in COVID-19 patients compared with controls
Analysis of the respiratory microbiota from the bronchoalveolar lavage liquid | at baseline and every 7 days during 28 days
  Alterations in respiratory microbiota composition (including virose, bacteria and fungi) in COVID-19 patients compared with controls
Serum inflammatory markers changes | at 28 days,
  Changes in blood, c-reactive protein, leucocyte, lymphocyte from baseline
Inflammatory markers changes | at 28 days,
  changes in Cytokine/ chemokine from baseline
Mortality | at 28 days,
  death
mechanical ventilation free days | at 28 days,
  Number of days alive without mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Saad Nseir, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHU Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No